CLINICAL TRIAL: NCT06761742
Title: An Artificial Intelligence Model for Accurate Diagnosis of Renal Tumors Based on Multi-phase Contrast-enhanced CT and Laboratory Tests: A Model Development and Multi-center Evaluation Study
Brief Title: Development of AI Model for Renal Tumor Diagnosis Using CT and Lab Tests
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Fudan University Pudong Medical Center (Unknown); Fudan University (Other); The Affiliated Hospital Of Southwest Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: DiagnosisModel_RenalTumor_AI
Record Dates: First submitted 2024-12-30; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Renal Tumors
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Training Set
- Validation Set
- Internal Test Set
- External Test Set

SUMMARY:
This multi-center retrospective study aims to develop a multimodal artificial intelligence diagnostic model using preoperative contrast-enhanced CT images and routine laboratory parameters from patients with renal tumors. The model is designed to assist clinicians in accurately predicting the pathological subtypes of renal tumors preoperatively, enabling detailed diagnoses and advancing precision medicine.

ELIGIBILITY:
Inclusion Criteria:

* Underwent renal tumor resection with a complete postoperative pathological report, and the pathological diagnosis is one of the following types: clear cell renal cell carcinoma, papillary renal cell carcinoma, chromophobe renal cell carcinoma, renal angiomyolipoma, or renal oncocytoma.
* Complete and available four-phase contrast-enhanced CT scans prior to surgery.
* Complete and available routine laboratory test results prior to surgery.

Exclusion Criteria:

* Incomplete CT data or poor image quality that affects diagnostic analysis.
* A time interval of more than three months between imaging or laboratory testing and pathological diagnosis.
* Patients diagnosed with fat-rich renal angiomyolipoma (AML).
* Pathological diagnosis indicating the coexistence of two or more pathological types of renal tumors.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients who underwent renal tumor resection at multiple centers, with complete preoperative imaging and laboratory data. Eligible participants include those with pathological diagnoses of clear cell renal cell carcinoma, papillary renal cell carcinoma, chromophobe renal cell carcinoma, renal angiomyolipoma, or renal oncocytoma. Patients with incomplete imaging data, poor-quality CT images, or coexistence of multiple pathological types of renal tumors were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 1922 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
postoperative pathological report | From the time of surgery to the release of the postoperative pathological report (typically within 2 weeks post-surgery).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to interested research partners upon reasonable request to Wei Zhai or Department of Urology, Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China.; the prerequisite for this is a data transfer agreement, approved by the legal departments of the requesting researcher and by all legal departments of the institutions that provided data for the study, and an ethics clearance.